CLINICAL TRIAL: NCT00231478
Title: A Randomized, Double-blind Study of 2 Dose Levels of Kytril on the Prevention of Post-operative Nausea and Vomiting in Pediatric Patients Undergoing Surgery With General Anesthesia
Brief Title: A Study of Kytril (Granisetron) in the Prevention of Post-Operative Nausea and Vomiting (PONV) in Pediatric Subjects Undergoing Tonsillectomy or Adenotonsillectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Clinical Trials, Study Director, Hoffmann-La Roche
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML16633
Record Dates: First submitted 2005-09-30; First posted 2005-10-04 (Estimated); Results first posted 2011-04-28 (Estimated); Last update posted 2018-03-27 (Actual); Status verified 2018-02

CONDITIONS: Post-Operative Nausea and Vomiting
MeSH Terms: conditions — Vomiting | interventions — Granisetron

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: granisetron
- 2 (Experimental)
  Interventions: Drug: granisetron

INTERVENTIONS:
Drug: granisetron — 20 micrograms intravenously (iv) 15 min prior to end of surgery
  Other Names: Kytril
  Arms: 1
Drug: granisetron — 40 micrograms intravenously (iv) 15 min prior to end of surgery
  Other Names: Kytril
  Arms: 2

SUMMARY:
This 2 arm study will evaluate the efficacy and safety of a single intravenous injection of Kytril in preventing postoperative nausea and vomiting (PONV) in children. Patients will be randomized to receive a single dose of either 20 micrograms or 40 micrograms Kytril intravenously (iv) 15 minutes prior to the end of surgery with general anesthesia for tonsillectomy or adenotonsillectomy. The anticipated time on study treatment is <3 months, and the planned sample size was 170 patients.

ELIGIBILITY:
Inclusion Criteria:

* males and females 2-16 years of age
* scheduled to undergo elective surgery for tonsillectomy or adenotonsillectomy requiring general anesthesia and endotracheal intubation
* scheduled for hospital admission for no longer than 24 hours

Exclusion Criteria:

* known allergy or other contraindication to the use of Kytril or any of its components
* known allergy to any other 5HT3 antagonist
* history of motion sickness or post-operative nausea or vomiting
* nausea or vomiting in the 24 hours prior to anesthesia

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 171 (Actual)
Dates: Start 2007-04; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (11):
- United States (11):
  - Fresno, California
  - Stanford, California
  - Hartford, Connecticut
  - Miami, Florida
  - Atlanta, Georgia
  - Indianapolis, Indiana
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Pittsburgh, Pennsylvania
  - Nashville, Tennessee
  - Dallas, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Granisetron 20 ug/kg: Drug: granisetron [Kytril], 20 micrograms intravenously (iv) 15 min prior to end of surgery
- Granisetron 40 ug/kg: Drug: granisetron [Kytril] , 40 micrograms intravenously (iv) 15 min prior to end of surgery
Period: Overall Study
Arm/Group | Granisetron 20 ug/kg | Granisetron 40 ug/kg
Started | 87 | 84
Completed | 79 | 78
Not Completed | 8 | 6
Not completed — Protocol Violation | 3 | 2
Not completed — Refused Treatment | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Adverse Event | 0 | 1
Not completed — Administrative | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Granisetron 20 ug/kg | Granisetron 40 ug/kg | Total
Number analyzed (Participants) | 70 | 73 | 143
Age, Continuous [Mean (Standard Deviation); unit: years] — The safety population was all evaluable population. The evaluable population consisted of 143 pediatric subjects from 2 to 16 years.
  years | 6.0 (3.37) | 6.2 (3.12) | 6.1 (3.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 43 | 65
  Male | 48 | 30 | 78

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With no Vomiting
Description: Number of patients with no vomiting is described as no emesis up to 2 hours after surgery
Time Frame: 0-2h after end of surgery (time of extubation)
Population: Evaluable Patients
Measure: Number; unit: participants
Arm/Group | Granisetron 20 ug/kg | Granisetron 40 ug/kg
Number analyzed (Participants) | 70 | 73
participants | 61 | 69

2. Secondary Outcome: Number of Patients With no Vomiting
Description: No vomiting describes no emesis during the first 24 hours
Time Frame: 0-24h after time of extubation
Population: Evaluable Patients
Measure: Number; unit: participants
Arm/Group | Granisetron 20 ug/kg | Granisetron 40 ug/kg
Number analyzed (Participants) | 70 | 73
participants | 49 | 50

3. Secondary Outcome: Time to First Vomiting Episode
Description: Time to first vomiting is described as the first event of emesis in hours. Subjects not having a vomiting episode are censored at the total length of time (in hours) between the time of extubation and time of the 24 hour follow-up.
Time Frame: 0-24h after time of extubation
Population: Evaluable Patients
Measure: Mean (Standard Error); unit: hours
Arm/Group | Granisetron 20 ug/kg | Granisetron 40 ug/kg
Number analyzed (Participants) | 70 | 73
hours | 18.0 (1.17) | 17.8 (1.12)

4. Secondary Outcome: Adverse Experiences
Description: The adverse events are captured in the AE and SAE section of this database
Time Frame: infusion to 15 days post treatment
Population: Eight of the 157 treated subjects (six and two in the 20- and 40-μg/kg dose groups,respectively) experienced a treatment-emergent serious adverse event up to 15 days after the treatment evaluation period.
Measure: Number; unit: Number of participants assessed
Arm/Group | Granisetron 20 ug/kg | Granisetron 40 ug/kg
Number analyzed (Participants) | 79 | 78
Number of participants assessed | 79 | 78

ADVERSE EVENTS:
Time Frame: Infusion to 15 days post treatment
Description: Eight of the 157 treated subjects (six and two in the 20- and 40-μg/kg dose groups,respectively) experienced a treatment-emergent serious adverse event up to 15 days after the treatment evaluation period.
Arm/Group | Granisetron 20 ug/kg | Granisetron 40 ug/kg
Serious Adverse Events (participants affected / at risk) | 6/79 | 2/78
Other Adverse Events (participants affected / at risk) | 6/79 | 4/78
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Granisetron 20 ug/kg (N=79) | Granisetron 40 ug/kg (N=78)
dehydration (General disorders) | 2 | 0
migraine (Vascular disorders) | 1 | 0
oral intake reduced (General disorders) | 1 | 1
post procedural haemorrhage (Surgical and medical procedures) | 2 | 1
oxygen saturation reduced (Metabolism and nutrition disorders) | 0 | 1
procedural pain (Surgical and medical procedures) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Granisetron 20 ug/kg (N=79) | Granisetron 40 ug/kg (N=78)
vomiting (Gastrointestinal disorders) | 6 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
"The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights."